CLINICAL TRIAL: NCT02288858
Title: A Multi-site, Double-blind, Placebo-controlled Clinical Study to Evaluate the Effects of Viviscal Oral Supplements When Used by Females With Self-perceived Thinning Hair
Brief Title: To Evaluate the Effects of Viviscal Oral Supplements When Used by Females With Self-perceived Thinning Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irish Response t/a Lifes2good (Industry)
Collaborators: Stephens & Associates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: L2G-Stephens-Viviscal
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Hair Thinning
Keywords: Hair thinning
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test product (Active Comparator): Viviscal Oral Supplement Tablets (as 512mg coated red-brown tablets in unbranded blister packs)
  Interventions: Dietary Supplement: Viviscal Oral Supplement Tablets
- Placebo (Placebo Comparator): Placebo Tablets (as 512 coated red-brown tablets in unbranded blister packs)
  Interventions: Dietary Supplement: Viviscal Oral Supplement Tablets

INTERVENTIONS:
Dietary Supplement: Viviscal Oral Supplement Tablets — Tablet (512 mg)

SUMMARY:
The purpose of this multi-site, double-blind, placebo-controlled clinical study, conducted for Lifes2Good, is to evaluate certain physiological effects of Viviscal Oral Supplement compared to a placebo in female subjects with self-perceived thinning hair associated with poor diet, stress, hormonal influences, or abnormal menstrual cycles.

Viviscal is an oral food supplement specifically designed to promote the quality of existing hair growth and/or to promote new hair re-growth for women suffering from temporary thinning hair. It does not contain hormones, drugs, or industry by-products. Viviscal has been marketed in Europe for over 15 years. The key ingredient is AminoMar C - a protein rich compound of marine extracts blended with soluble silica and fortified with Vitamin C. Viviscal provides essential nutrients to nourish hair naturally from within. Viviscal works over several months of use to improve the appearance of thinning hair.

DETAILED DESCRIPTION:
The purpose of this multi-site, double-blind, placebo-controlled clinical study, conducted for Lifes2Good, is to evaluate certain physiological effects of Viviscal Oral Supplement compared to a placebo in female subjects with self-perceived thinning hair associated with poor diet, stress, hormonal influences, or abnormal menstrual cycles. A total of 72 female subjects (36 subjects at the Dallas Research Center and 36 subjects at the Colorado Research Center) completed the study.

At day 0, prior to clinical procedures, subjects were assigned to 1 of the 2 treatment groups, Viviscal Oral Supplement or Placebo Tablets, based on the completely randomized study design that was generated with no input of subject information and conditions. During the course of the study, subjects consumed 1 tablet (512 mg) 3 times per day of the assigned test material, Viviscal Oral Supplement or Placebo Tablets, with water after food.

Clinical evaluations were conducted at visit 1 (day 0), visit 2 (day 2), visit 3 (3 months ± 2 weeks), visit 4 (2 days after visit 3), visit 5 (6 months ± 2 weeks), and visit 6 (2 days after visit 5). Subjects participated in the following procedures at the indicated time points:

* Scalp Examination At day 0, each subject's scalp was examined by the Sub-Investigator to rule out any confounding scalp conditions.
* Physical Examination A qualified nurse/nurse practitioner performed a basic physical examination of each subject at day 0, 3 months±2 weeks, and 6 months±2 weeks. The physical examination included a basic body systems overview, vital signs (blood pressure and pulse), respiration rate, temperature, weight, and height. Additionally, at the Colorado Research Center, the Sub-Investigator and qualified nurse practitioner examined each subject's scalp.
* Test Site Selection and Preparation At day 0, the examining Sub-Investigator selected a target area on each subject's scalp. To prepare the target areas for digital photography, subjects underwent shaving of the target areas at day 0, 3 months±2 weeks, and 6 months±2 weeks. Hair dyeing of the target areas was performed at day 0 and (if fading had occurred) at day 2, 3 months±2 weeks, 2 days after visit 3, 6 months±2 weeks, and 2 days after visit 5. Subjects underwent demarcation of the target areas with a small black dot tattoo at day 0 and (if fading had occurred) at 3 months±2 weeks and 6 months±2 weeks. For post-day 0 time points, tattooing procedures (if needed) were performed after the photography procedures.
* Digital Photography Macro photographs were captured of each subject's target area selected by the Sub-Investigator at all study visits.
* Shed Hair Collection Procedures At day 2, 2 days after visit 3, 2 days after visit 5, a clinician shampooed each subject's hair in a normal washing manner over a sink with securely fastened cheesecloth positioned to catch any hairs that were shed from the scalp. A clinician gently combed through the hair and rinsed any shed hairs from the comb onto the cheesecloth. Shed hairs found in the cheesecloth were counted and recorded.
* Questionnaire Each subject completed a quality of life questionnaire at baseline (day 0), 2 days after visit 3 and 2 days after visit 5 and a consumer questionnaire at 2 days after visit 3 and 2 days after visit 5.
* Daily Diary During the course of the study, subjects completed a daily diary to record product application times, any comments, and responses to a weekly question regarding their hair loss.
* Interviews At day 0, a portion of the subjects (at the Dallas Research Center) was selected to be interviewed and filmed. Film interviews were conducted for the pre-selected subjects at day 2 and 2 days after visit 5.

ELIGIBILITY:
Inclusion Criteria:

1. Females, ages 21-55 years of age.
2. Clinically-determined general good health as determined by responses to the initial paperwork.
3. Females with self-perceived thinning hair associated with poor diet, stress, hormone influences or abnormal menstrual cycle.
4. Females willing to maintain their normal hair shampooing frequency.
5. Females willing to add the provided oral supplement to their current daily routine.
6. Females willing to not substantially change their current diet, medications, or exercise routines for the duration of the study. If a subject receives physician guidance during the study to change diet, medications, or exercise routine, the subject will need to notify the clinic as soon as possible.
7. Females willing to undergo a brief physical exam to include height, weight, blood pressure, pulse, general physical findings and a scalp exam. The physical exam will occur at Visits 1, 3, and 5.
8. Females willing to have a small dot tattoo applied to the scalp, a small area of hair shaved (approximately 1 cm2) to approximately 1 mm in length, remaining hair in that small area dyed black, and to have photographs performed. If the dot tattoo fades substantially by Visit 3, it may need to be re-inked.
9. Females willing to wash their hair at the testing facility at Visits 2, 4 and 6 with the provided normal shampoo. Subjects may bring their own conditioner to use after shampooing.
10. Individuals with Fitzpatrick I-III photo skin types, (Fitzpatrick IV may be enrolled at the discretion of the clinical investigator).
11. Willingness to maintain a consistent haircut and hair color throughout the 6 month study period.

Exclusion Criteria:

1. Females with a known history of intolerance or allergy to fish, seafood or acerola.
2. Individuals with any known allergy or sensitivity to any shampoo/conditioner.
3. Females who are nursing, pregnant, planning to become pregnant during the study.
4. Females who are participating on any clinical research study at Stephens or at another research center or doctor's office.
5. Females who have recently (within the last 6 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (6 months or longer) in order to be eligible for the study.
6. Females currently using the HairMax light treatment to treat thinning hair.
7. Females who have regularly used Rogaine (Minoxidil) or Nizoral/Ketoconazole within the last 3 months.
8. Females who have used prescription drugs known to affect the hair growth cycle within, 6 months (e.g., hormone-based birth control for less than 6 months).
9. Females suffering from other hair loss disorders, such as alopecia areata, scarring alopecia or androgenetic alopecia.
10. Females who have had hair transplants within 6 months of study start.
11. Individuals with self-reported uncontrolled diseases (i.e. diabetes, hypertension, hyperthyroidism, hypothyroidism, etc. Medical conditions that are under control with or without treatment will be considered on an individual basis by the Investigators.
12. Females with self-reported active hepatitis, immune deficiency, HIV or autoimmune disease.
13. Females having a known active dermatologic condition which, in the opinion of the examining Investigator, might place the subject at a greater risk or interfere with clinical evaluations (e.g., seborrheic dermatitis, psoriasis, atopic dermatitis, advanced skin cancer, etc.)

Ages: 24 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Hair shedding rate | 6 months
  The numbers of scalp hairs shed at month 3 and month 6 when compared with baseline values.
Hair fiber diameter | 6 months
  Mean vellus hair width change

SECONDARY OUTCOMES:
Quality of life questionnaires | 6 months
  Quality of life questionnaires relating to perception of quality of hair growth and their wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald L Rizer, PhD, Principal Investigator — Stephens & Associates, Inc.
Locations (1):
- Stephens Associates Inc., Richardson, Texas, United States